CLINICAL TRIAL: NCT00652886
Title: Compare the Relative Bioavailability of Oxandrolone 10mg Tablets With That of OXANDRIN 10 mg Tablets Following a Single Oral Dose(1*10 mg Tablet) in Healthy, Adult Subjects Under Fasting Conditions.
Brief Title: Bioavailability Study of Oxandrolone Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Cetero Research, San Antonio (Network)
Responsible Party: Dr. Alfred Elvin, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B053205
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: To Determine the Bioequivalence Under Fasting Conditions
Keywords: Bioequivalence, Oxandrolone,fasting
MeSH Terms: conditions — Fasting | interventions — Oxandrolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received Kali's products under fasting conditions
  Interventions: Drug: Oxandrolone
- B (Active Comparator): Subjects received BTG products under fasting conditions
  Interventions: Drug: Oxandrin

INTERVENTIONS:
Drug: Oxandrolone — Tablets, 10mg, single-dose
  Other Names: Oxandrin
  Arms: A
Drug: Oxandrin — tablets, 10mg, single-dose
  Other Names: Oxandrolone
  Arms: B

SUMMARY:
-To compare the single dose bioavailability of Kali and BTG

DETAILED DESCRIPTION:
-To compare the bioavailability of Oxandrolone 10mg tablets with that of OXANDRIN 10mg tablets following a single -dose in healthy, adult subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject at least 18 years of age, may be male or they may be female who are unable to bear children.
* Each subject shall be given a general physical examination within 28days of the initiation study.
* At the end of the study, the subjects will have an exit evaluation consisting of interim history, global evaluation, and clinical laboratory measurements.
* Each female subject will be given a serum test as part of the pregnancy study screening process.
* Clinical laboratory measurements will include Hematology, Clinical Chemistry, Urine Analysis, HIV Screen,hepatitis-B, C screen and Drugs of abuse Screen

Exclusion Criteria:

* Subjects with a history of alcoholism or drug addiction(during past 2 years), or serious gastrointestinal, renal hepatic or cardiovascular disease, tuberculosis, epilepsy. asthma, diabetes, psychosis or glaucoma will not be eligible for thsi study.
* Subjects with any history of breast or prostate cancer will not be eligible to participate in this study.
* Subjects who have a history of allergic response to the class of drug being tested will be excluded from the study.
* Subjects found to have urine/saliva concentration of any of the tested drugs will not be allowed to participate.
* Subjects who have taken any investigational drug within thirty days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are not able to bear children will not be allowed to participate.
* Female subjects with positive or inconclusive results will be withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-03; Primary Completion 2005-03 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Steve Herrmann, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc, Saint Charles, Missouri, United States